CLINICAL TRIAL: NCT03561571
Title: Composition of Triglyceride Rich Lipoproteins and Platelet Activation in Type 2 Diabetic Women
Brief Title: Triglyceride Rich Lipoproteins and Platelet Activation in Type 2 Diabetes
Acronym: COMPLETE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL18_0326
Record Dates: First submitted 2018-05-25; First posted 2018-06-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2019-08

CONDITIONS: Type2 Diabetes
Keywords: chylomicrons; Very Low Density Lipoprotein; saturated fat; platelet function; type 2 diabetes; post prandial phase
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butter based breakfast (Active Comparator)
  Interventions: Other: butter based breakfast
- Chocolate spread based breakfast (Active Comparator)
  Interventions: Other: Chocolate spread based breakfast

INTERVENTIONS:
Other: butter based breakfast — ingestion of proteins : 5 g, lipids 20 g, glucides 57 g
  Arms: Butter based breakfast
Other: Chocolate spread based breakfast — ingestion of proteins 7 g, lipids 20 g, glucides 56 g
  Arms: Chocolate spread based breakfast

SUMMARY:
To investigate in vitro the effect of triglyceride rich lipoproteins (TGRL) obtained in type 2 diabetic women in the fasting state and following a randomized isocaloric lipid rich breakfast on control human platelets

Randomized Comparison of butter versus chocolate spread in 2 groups of 15 patients

ELIGIBILITY:
Inclusion Criteria:

* Menopausal women
* HbA1c ≥6,5 ou ≤10%
* 27 ≤ BMI ≤40 kg/m2

Exclusion Criteria:

* Insulin therapy
* fibrates or Omega 3 fatty acids supplements
* Hormonal replacement therapy of menopause
* Glycemia > 16 mmol/l
* Alcohol abuse (≥3 Unit/day)
* Special dietary habits
* History of bariatric surgery

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
fasting thromboxane B2 concentration | Hour 0
  ex vivo experiment : TGRL obtained by preparative Unesterified cholesterol (UC) incubated with control human platelets
after breakfast thromboxane B2 concentration | 4 hours
  ex vivo experiment : TGRL obtained by preparative Unesterified cholesterol (UC) incubated with control human platelets

SECONDARY OUTCOMES:
measurement of fasting platelet activation by turbidimetric method | Hour 0
measurement of post prandial platelet activation by turbidimetric method | 4 Hours
fasting lipidomic composition of triglyceride rich lipoproteins | Hour 0
  Characterization and comparison of LRT lipidomics in fasting DT2 patients and following the ingestion of a high-fat breakfast according to their source (short and medium chain fatty acids (butter) versus palmitic acid (palm oil present in spreads).
post prandial lipidomic composition of triglyceride rich lipoproteins | 4 Hours
  Characterization and comparison of LRT lipidomics in fasting DT2 patients and following the ingestion of a high-fat breakfast according to their source (short and medium chain fatty acids (butter) versus palmitic acid (palm oil present in spreads).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel - department of endocrinology, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Boulet MM, Cheillan D, Di Filippo M, Lelekov-Boissard T, Buisson C, Lambert-Porcheron S, Nazare JA, Tressou J, Michalski MC, Calzada C, Moulin P. Postprandial Triglyceride-Rich Lipoproteins from Type 2 Diabetic Women Stimulate Platelet Activation Regardless of the Fat Source in the Meal. Mol Nutr Food Res. 2020 Oct;64(19):e2000694. doi: 10.1002/mnfr.202000694. Epub 2020 Sep 9. PMID 32844550